CLINICAL TRIAL: NCT03873649
Title: CD4 T-cell Immunephenotype in Hypersensitivity Pneumonitis
Brief Title: Immune Response in Hypersensitivity Pneumonitis
Status: Completed | Type: Observational
Sponsor: Nabeel Hamzeh (Other)
Collaborators: National Jewish Health (Other)
Responsible Party: Sponsor-Investigator, Nabeel Hamzeh, Associate Professor of Medicine, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201805937
Record Dates: First submitted 2019-02-27; First posted 2019-03-13 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Hypersensitivity Pneumonitis
MeSH Terms: conditions — Alveolitis, Extrinsic Allergic | interventions — Bronchoscopy; Therapeutic Irrigation; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with subacute or chronic hypersensitivity pneumonitis: Procedures that each subject will undergo include:
  1. Chest CT scan to determine extent of disease.
  2. Pulmonary function testing to determine severity of disease.
  3. Bronchoscopy with lavage.
  4. Venipuncture.
  Interventions: Other: Bronchoscopy with lavage
- Healthy Controls: Inclusion:
  1. Adult between the ages of 18 and 80 years old.
  2. Non-smoker or previous smoker quit >6months ago.
  3. Able to understand the consent process and procedures involved in the study.
  Exclusion:
  1. Unable to understand the consent process or procedures involved in the study.
  2. Pregnancy.
  3. Suspicion of current infection or within the past 3 months.
  4. Bleeding disorder or on anti-coagulants other than aspirin.
  5. Any co-morbid condition that increases risk of bronchoscopy including but not limited to cardiac disease, uncontrolled hypertension, uncontrolled diabetes and/or morbid obesity.
  Interventions: Other: Bronchoscopy with lavage

INTERVENTIONS:
Other: Bronchoscopy with lavage — Bronchoscopy will be performed according to standard clinical procedures. Bronchoscopy will be performed under conscious sedation with continuous cardiopulmonary monitoring and the subject's upper airway will be anesthetized with topical lidocaine. The bronchoscope will be passed through the naris or mouth to the upper airway and then into the lower airway. 360cc of sterile saline will be instilled into 2 sub-segments by instilling and aspirating 3 aliquots of 60cc sequentially into each sub-segment.
  Venipuncture to obtain peripheral blood mononuclear cells (PBMCs) for the proposed assays.
  Cells collected will be analyzed for various T-cell subsets and gene expression to help determine the type of immune response.
  Other Names: blood draw

SUMMARY:
Hypersensitivity pneumonitis (HP) is an inflammatory lung disease that is caused by exposure of susceptible individuals to organic materials in the environment. It is also known by various names depending on the exposure and some of these names include farmer's lung, pigeon breeder's lung, hot tub lung to name a few. HP can cause lung scarring that impairs breathing and oxygenation. Early detection and avoidance of triggers can stop and reverse the disease but a significant number of patients continue to have active disease requiring treatment in spite of avoiding the trigger. The current choice of therapies is based on clinical experience and not on rigorous clinical trials. Not fully understanding the type of inflammation that is seen in HP and the cells involved in this inflammatory response limits health care providers' ability to choose drugs to study in HP that can stop the inflammation and limit scar formation. The goal of the investigators' study is to better understand the type of cells that are involved in the inflammatory response in the lungs of HP patients and what drives these cells to be active. By better understanding the type of cells and what drives them, health care providers can begin to choose and study drugs that can limit the inflammation and subsequent scarring. The investigators' will recruit HP patients and with their consent perform a scope of the lungs (bronchoscopy) with a limited lung wash to get the inflamed cells out of the lungs to further study them in the lab. The investigators' study will provide us with preliminary results to guide us in performing a more detailed study in the future to better understand the disease.

DETAILED DESCRIPTION:
Hypersensitivity pneumonitis (HP) is a granulomatous lung disorder triggered by exposure to one of a multitude of organic antigens. Incidence rates of HP vary by geography, season and population studied but it is estimated to be the third most common interstitial lung disease with an estimated prevalence rate in the USA of 420-3000/100,0002. HP accounts for at least 7.5% of ILD related lung transplant. Exposure to an antigen in a susceptible host induces an inflammatory response with the subsequent formation of poorly formed granulomas that impact gas exchange which clinically manifests as shortness of breath, hypoxia and radiographic changes. HP can present acutely, subacutely or chronically depending on the duration of symptoms and radiographic changes. Radiographic manifestations of HP include ground-glass changes, centrilobular nodules, air trapping known as mosaic pattern, fibrosis, emphysema, or more frequently a combination of these. The cornerstone of management is identification and avoidance of the inciting agent which is effective if accomplished early in the disease process.

Although detection and avoidance of possible triggers can attenuate or reverse the disease, a significant number of patients continue to have active and/or progressive disease requiring chronic immunosuppressive therapy. Standard of care for IS therapy is corticosteroids and azathioprine but this is based on clinical experience and not based on randomized clinical trials(ref). The efficacy of this regimen is not known and patients develop persistent or progressive disease in spite of aggressive therapy leading to end stage lung disease necessitating lung transplantation or ending with death. To date, there are no randomized trials for immunosuppressive therapies and no reports of the use of biological agents in HP. The lack of studies is partially due to the lack of a thorough understanding of the immune response in HP especially in patient based studies that focus at the site of disease activity, the lungs.

The immunological response and pathways leading to this response have not been fully investigated especially in humans. The Th17 pathway has been implicated in disease pathogenesis and T-regulatory cell dysfunction has been described although studies in humans are limited. Recent work in sarcoidosis, a granulomatous lung disease, has shown that Th17.1 cells play a potential important role in granuloma immunopathogenesis. Through an R01 mechanism, the investigators are currently investigating the role of T-cell skewing and associated gene expression in sarcoidosis that is associated with progressive disease vs stable disease and the investigators are investigating its impact on disease course.

This gap in knowledge in HP has limited the choice and study of immunomodulatory agents in HP and especially biological agents in the treatment of persistent and progressive disease. To narrow this knowledge gap, the investigators propose conducting a study to investigate the lung CD4+ T-cell immunophenotype and CD4+ T-cell gene expression in HP to enhance the investigators' understanding of the immune response in HP and the pathways involved in the immune response which would enable the investigators to further pursue guided therapeutic trials in subacute and chronic HP.

ELIGIBILITY:
Inclusion:

1. Adult between the ages of 18 and 80 years old.
2. Non-smoker or previous smoker quit >6months ago.
3. Radiological findings compatible with sub-acute or chronic HP4.
4. Histopathological findings compatible with sub-acute or chronic HP4.
5. Able to understand the consent process and procedures involved in the study.

Exclusion:

1. Unable to understand the consent process or procedures involved in the study.
2. End-stage lung disease defined as predominantly honeycombing on chest CT and/or FVC<60% and/or DLCO <30%.
3. Requiring high oxygen needs >4L.
4. Pregnancy.
5. Treated with a biological agent within the past 6 months.
6. Suspicion of current infection or within the past 3 months.
7. Bleeding disorder or on anti-coagulants other than aspirin.
8. Any co-morbid condition that increases risk of bronchoscopy including but not limited to cardiac disease, uncontrolled hypertension, uncontrolled diabetes and/or morbid obesity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypersensitivity Pneumonitis patients with confirmed subacute and chronic HP based on compatible radiological and pathological findings will be eligible for recruitment
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
T-cell subtypes | outcomes will be assessed after recruitment is complete in 2 years.
  T-cell subtypes will be determined by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Nabeel Hamzeh, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No